CLINICAL TRIAL: NCT06077188
Title: Erciyes University
Brief Title: EFFECT of CHEWING GUM on CONTROLLING NAUSEA/VOMITING and THIRST in PATIENTS with ACUTE PANCREATITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Teaching staff, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Thirstgum
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-02

CONDITIONS: Acute Pancreatitis; Thirst
Keywords: Acute Pancreatitis; Thirst; nouse; vomiting
MeSH Terms: conditions — Pancreatitis; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Gum group
- Control group (No Intervention)

INTERVENTIONS:
Other: Gum group — Group chewing gum with xylitol
  Arms: intervention group

SUMMARY:
Nausea and vomiting are one of the most common symptoms in acute pancreatitis. In addition to pharmacological methods for nausea and vomiting, non-pharmacological methods can also be used. Among these, anticipatory nausea and vomiting can be prevented by behaviors aimed at distracting attention. This study will be conducted to evaluate the effect of chewing gum on the severity of nausea-vomiting and thirst in patients with acute pancreatitis. The study will be conducted with a total of 60 patients, 30 intervention and 30 control.

Patients in the intervention group will chew xylitol gum five times a day for three days. The patients' thirst and nausea and vomiting conditions will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with acute pancreatitis,

  * Without total dental prosthesis,
  * Without salivary gland infection,
  * Those who have not had salivary gland surgery,
  * No difficulty in chewing,
  * Not receiving oxygen therapy,
  * Able to answer all questions and be communicativ

Exclusion Criteria:

* Those with diabetes,
* Does not like chewing gum,
* Receiving radiotherapy or chemotherapy,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Thirst Severity -Visual Analog Scale | Apply in the morning of the 1st day after application
  Visual Analog Scale is a 10 cm long scale that evaluates the severity of thirst.

SECONDARY OUTCOMES:
Rhodes Nausea, Vomiting and Retching Index | Apply in the morning of the 1st day after application
  It is an eight-item scale that measures the number and severity of patients' nausea, vomiting and retching in the last 24 hours.
Rhodes Nausea, Vomiting and Retching Index ( | Apply in the morning of the 1st day after application
  It is an eight-item scale that measures the number and severity of patients' nausea, vomiting and retching in the last 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hospital, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Jensdottir T, Buchwald C, Nauntofte B, Hansen HS, Bardow A. Saliva in relation to dental erosion before and after radiotherapy. Acta Odontol Scand. 2013 May-Jul;71(3-4):1008-13. doi: 10.3109/00016357.2012.741704. Epub 2012 Nov 21. PMID 23167908
- [Background] Oyetola EO, Owotade FJ, Agbelusi GA, Fatusi OA, Sanusi AA. Oral findings in chronic kidney disease: implications for management in developing countries. BMC Oral Health. 2015 Feb 20;15:24. doi: 10.1186/s12903-015-0004-z. PMID 25888327
- [Background] Silva AC, Aprile LR, Dantas RO. EFFECT OF GUM CHEWING ON AIR SWALLOWING, SALIVA SWALLOWING AND BELCHING. Arq Gastroenterol. 2015 Jul-Sep;52(3):190-4. doi: 10.1590/S0004-28032015000300007. PMID 26486285
- [Background] Honarmand M, Farhad-Mollashahi L, Nakhaee A, Sargolzaie F. Oral manifestation and salivary changes in renal patients undergoing hemodialysis. J Clin Exp Dent. 2017 Feb 1;9(2):e207-e210. doi: 10.4317/jced.53215. eCollection 2017 Feb. PMID 28210437